CLINICAL TRIAL: NCT07126847
Title: Evaluation of the Success of POCUS Usage in Addition to STONE Criteria in Diagnosing Nephrolithiasis and Predicting Readmission Within One Month in Patients Presenting to the Emergency Department With Suspected Nephrolithiasis
Brief Title: Use of POCUS and STONE Criteria Together in the Diagnosis of Nephrolithiasis
Acronym: POCUS
Status: Active, not recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-10
Record Dates: First submitted 2024-03-27; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Renal Colic; Stone, Kidney; Hydronephrosis; Nephrolithiasis
Keywords: POCUS; STONE; Renal Colic; Nephrolithiasis
MeSH Terms: conditions — Renal Colic; Kidney Calculi; Hydronephrosis; Nephrolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Renal Ultrasonography — To investigate the primary and secondary signs of stones with ultrasound and to additionally use the Stone criteria in patients with suspected nephrolithiasis.
  Other Names: STONE criteria

SUMMARY:
Patients presenting to the emergency department with symptoms suggestive of renal colic will be included in the study at Kocaeli City Hospital's emergency department. Patients with nephrolithiasis considered among the preliminary diagnoses will be enrolled in the study; demographic data, vital signs, and physical examination findings will be recorded on pre-prepared standard data forms.

STONE criteria scores will be calculated by emergency assistants, and bedside ultrasound will be performed for patients. Ultrasonographic findings suggestive of renal colic, such as hydronephrosis, the presence of primary stones, acoustic shadowing of the stone, the presence of twinkle artifact, presence of jet flow, and presence of bladder debris, will be evaluated, and the obtained data will be recorded on the standard data form by the performing assistant physician. In patients where computed tomography, which is the gold standard for detecting stone presence without intervention, is deemed appropriate without any intervention to the primary examining physician, the computed tomography results and ultrasound findings will be compared.

The study aims to evaluate the effectiveness of bedside ultrasound application in diagnosing stone presence in patients, its success in predicting re-admission to the hospital within 1 month, its success in predicting possible alternative diagnoses and complications, in addition to the stone criteria applied in the patients.

DETAILED DESCRIPTION:
Our study is a prospective study that will be conducted in the Emergency Medicine Clinic of Kocaeli City Hospital. Patients aged 18 and above who present to the emergency department of Kocaeli City Hospital with symptoms suggestive of renal colic will be included in the study if they volunteer. After examination by a resident physician working in the emergency department, patients for whom nephrolithiasis is considered among the preliminary diagnoses will be notified to the principal investigators. After obtaining written consent, demographic data, vital signs, and physical examination findings will be recorded on previously prepared standard data forms.

Patients scoring 8 points or higher according to the STONE criteria based on history, physical examination, and laboratory results will undergo bedside ultrasound. The ultrasound will be performed by 4 resident physicians with a basic ultrasound course certificate from the Turkish Emergency Medicine Association, who have 2 years of experience. The bedside urinary ultrasound will be performed using the 'Esaote Mylab Gamma® device (Genoa, Italy)' ultrasound machine with the 'Esaote AC2541 curved array (1-8 MHz) probe (Genoa, Italy)' while the patient is in the supine position.

During renal ultrasound, the convex ultrasound probe will be placed in the right upper quadrant of the patient, intersecting the right lower intercostal area and the mid-axillary line. In the left upper quadrant, the probe will be placed in the lower intercostal area along the posterior axillary line. The ultrasound probe will be positioned longitudinally with the indicator pointing towards the patient's head. Subsequently, the same area will be imaged transversely with the indicator pointing towards the patient's right.

In these sections, images of the kidneys will be evaluated for the presence of hydronephrosis, the degree of expansion of pelvic-calyceal structures, stone size, kidney dimensions, parenchymal echogenicity, and the presence of primary stones or acoustic shadowing from stones. Then, from the suprapubic region, the probe will be positioned transversely and longitudinally, sequentially showing the patient's right and head; the presence of globules in the bladder, bladder dimensions, the presence of stones, and the degree of jet flow at the junction of the ureters with the bladder will be assessed using color frequency mode (CFM). The presence of twinkling artifacts with color frequency mode (CFM) will be evaluated when a stone is suspected. The data obtained will be recorded on the study form by the resident physician performing the ultrasound. The recorded data will later be compared with the gold standard diagnostic method, computed tomography routinely performed in patients with nephrolithiasis, for effectiveness.

ELIGIBILITY:
Inclusion Criteria:

- All volunteer patients

Exclusion Criteria:

* Pregnant patients,
* Patients for whom the clinician does not give an indication for computed tomography,
* Patients with a previous history of nephrectomy and kidney transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteer patients over the age of 18 who applied to the emergency department of Kocaeli City Hospital with renal colic will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Nephrolithiasis diagnostic accuracy | 2 year
  Adding bedside focused ultrasonography to the STONE criteria increases diagnostic accuracy in patients presenting to the emergency department with a preliminary diagnosis of nephrolithiasis.

SECONDARY OUTCOMES:
Predicting the possible complications | 2 year
  The success of using POCUS in predicting possible complications in patients with nephrolithiasis.
Readmission to hospital. | 1 month
  Predicting hospital readmission rate within 1 month in patients with nephrolithiasis.

CONTACTS AND LOCATIONS:
Overall Officials: Asım Enes Özbek, Study Director — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rosen's Emergency Medicine: Concepts and Clinical Practice 10th Edition-June 13, 2022 Authors: Ron Walls, Robert Hockberger, Marianne Gausche-Hill, Timothy B. Erickson, Susan R. Wilcox
- [Background] Teichman JM, Long RD, Hulbert JC. Long-term renal fate and prognosis after staghorn calculus management. J Urol. 1995 May;153(5):1403-7. PMID 7714951
- [Background] Preminger GM, Tiselius HG, Assimos DG, Alken P, Buck C, Gallucci M, Knoll T, Lingeman JE, Nakada SY, Pearle MS, Sarica K, Turk C, Wolf JS Jr; EAU/AUA Nephrolithiasis Guideline Panel. 2007 guideline for the management of ureteral calculi. J Urol. 2007 Dec;178(6):2418-34. doi: 10.1016/j.juro.2007.09.107. No abstract available. PMID 17993340
- [Background] Westphalen AC, Hsia RY, Maselli JH, Wang R, Gonzales R. Radiological imaging of patients with suspected urinary tract stones: national trends, diagnoses, and predictors. Acad Emerg Med. 2011 Jul;18(7):699-707. doi: 10.1111/j.1553-2712.2011.01103.x. PMID 21762233
- [Background] Berrington de Gonzalez A, Mahesh M, Kim KP, Bhargavan M, Lewis R, Mettler F, Land C. Projected cancer risks from computed tomographic scans performed in the United States in 2007. Arch Intern Med. 2009 Dec 14;169(22):2071-7. doi: 10.1001/archinternmed.2009.440. PMID 20008689
- [Background] Moore CL, Carpenter CR, Heilbrun ML, Klauer K, Krambeck AC, Moreno C, Remer EM, Scales C, Shaw MM, Sternberg KM. Imaging in Suspected Renal Colic: Systematic Review of the Literature and Multispecialty Consensus. J Urol. 2019 Sep;202(3):475-483. doi: 10.1097/JU.0000000000000342. Epub 2019 Aug 8. PMID 31412438
- [Background] Smith-Bindman R, Aubin C, Bailitz J, Bengiamin RN, Camargo CA Jr, Corbo J, Dean AJ, Goldstein RB, Griffey RT, Jay GD, Kang TL, Kriesel DR, Ma OJ, Mallin M, Manson W, Melnikow J, Miglioretti DL, Miller SK, Mills LD, Miner JR, Moghadassi M, Noble VE, Press GM, Stoller ML, Valencia VE, Wang J, Wang RC, Cummings SR. Ultrasonography versus computed tomography for suspected nephrolithiasis. N Engl J Med. 2014 Sep 18;371(12):1100-10. doi: 10.1056/NEJMoa1404446. PMID 25229916
- [Background] Moore CL, Bomann S, Daniels B, Luty S, Molinaro A, Singh D, Gross CP. Derivation and validation of a clinical prediction rule for uncomplicated ureteral stone--the STONE score: retrospective and prospective observational cohort studies. BMJ. 2014 Mar 26;348:g2191. doi: 10.1136/bmj.g2191. PMID 24671981